CLINICAL TRIAL: NCT06904612
Title: Micronutrient-fortified Iodized Salt and Serum Concentrations of Folate, B12 and Iron in Reproductive-aged Women of Rural India
Brief Title: Using Iodized Salt to Improve Serum Folate, B12 and Iron Levels
Status: Completed | Type: Observational
Sponsor: Hydrocephalus and Neuroscience Institute (Other)
Collaborators: Andhra Medical College (Other Government)
Responsible Party: Sponsor
Other Study IDs: CT06174883; 191/IEC AMC/MAY 2021 (Other: Andhra Medical College Institutional Ethics Committee)
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Neural Tube Defects; Folic Acid Deficiency; Spina Bifida; Anencephaly-Spina Bifida; B12 Deficiency Vitamin; Anemia; Iron Deficiency Anaemia Due to Dietary Causes
Keywords: Micronutrient deficiency; Food fortification; dietary salt; India; Folic acid; Neural tube defects; Spina Bifida; anencephaly; anemia; B12 deficiency
MeSH Terms: conditions — Neural Tube Defects; Folic Acid Deficiency; Spinal Dysraphism; Neural tube defects X-linked; Vitamin B 12 Deficiency; Anemia; Anencephaly

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Micronutrient fortified iodized salt — addition of folic acid, B12 and iron to iodized salt to be consumed daily and assess rise in serum levels.

SUMMARY:
Question: How effective is fortified iodized salt in increasing serum concentrations of folate, B12 and iron among non-pregnant and non-lactating women of reproductive age?

Hypothesis: Micronutrient fortified iodized salt can increase serum levels (of folate, B12 and iron) and serve as a policy consideration in salt fortification with both iodine and other micronutrients to reduce serious and fatal birth defects.

DETAILED DESCRIPTION:
Salt is an ideal vehicle for fortification because its universal consumption and often centrally processed with established distribution channels. Over 70% of households globally have access to iodized salt. Considering the success of salt iodization, it is logical to use the existing infrastructure to provide folic acid and other micronutrients (such as B12 and iron) through this dietary mechanism.

AIM:To assess increase in blood concentrations of folate, B12 and iron among women of reproductive age who consume micronutrient-fortified iodized salt for 3 months.

OBJECTIVES :

1. To examine the effect of consumption of iodized salt fortified with folic acid, B12 and iron on serum/plasma concentrations among women of reproductive age.
2. To assess acceptance of study salt for daily use during 3 months of consumption.

ELIGIBILITY:
Inclusion Criteria: • Willing to voluntarily participate in the study

* Can comprehend and comply with study requirements
* Aged between 18 and 45 years.
* No documented issues with child bearing potential
* Resident of the area of study for duration of study.
* Consume only study salt during study

Exclusion Criteria:

* Taking multivitamins or micronutrient supplements during study
* Pregnant or lactating at recruitment or during study
* Co-morbidities such as Malabsorption disorders, severe anemia (Hgb <8.0 g/dL), uncontrolled hypertension, (SBP ≥140 mm Hg or DBP ≥90 mm Hg), HIV, active TB or malaria infection
* History of prior SBA delivery
* Pre-existing medical conditions (i.e., cancer or need for regular medications)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women of childbearing age
Study Population: Women of childbearing age who are non-lactating and willing to consume the study salt for the duration were recruited for voluntary participation into the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Measure changes in median serum folate, B12 and iron levels between baseline and study endpoint | 2-6 months
  evaluate blood levels pre- and post-intake of study salt (fortified with folic acid, B12 and iron)

CONTACTS AND LOCATIONS:
Overall Officials: Jogi Pattisapu, MD, Principal Investigator — Pediatric Neurosurgery
Locations (2):
- Pediatric Neurosurgery, Orlando, Florida, United States
- Andhra Medical College, Visakhapatnam, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided
redacted information will be made available upon request.